CLINICAL TRIAL: NCT03422900
Title: Influence of Two Enteral Nutrition Formulas on Hyperglycemia and Morbidity in Patients with Stroke
Brief Title: Hyperglycemia in Patients with Stroke and Indication of Enteral Nutrition
Acronym: GlyENStroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endocrinology and Clinical Nutrition Research Center, Spain (Other)
Responsible Party: Principal Investigator, Daniel de Luis Roman, Profesor Doctor, Endocrinology and Clinical Nutrition Research Center, Spain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASVE-NM-17-315
Record Dates: First submitted 2017-12-10; First posted 2018-02-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Hyperglycaemia (Non Diabetic); Enteral Feeding Intolerance; Stroke
MeSH Terms: conditions — Hyperglycemia; Stroke | interventions — (4-(4,5-dihydro-1H-imidazol-2-yl)amino)benzoic acid

STUDY DESIGN:
Intervention Model Description: Comparison of two formulas of enteral nutrition (diabetes-specific enteral formula (lower glycemic index and presence of soluble and insoluble fiber) compared to an standard formula (isocaloric and isonitrogenated formula without fiber)) in patients without diabetes mellitus admitted due to stroke and with indication of nutritional support by nasogastric tube
Who Masked: Participant, Care Provider
Masking Description: cover label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Specific Diabetes Formula (Experimental): Diabetes-Specific Enteral Formula:
  * Caloric density: 1,0 kcal/ml
  * Energy: 100 kcal
  * Carbohydrates: 10,1 g/100 ml;
  * Fat: 4,5 g/100 ml
  * Prot: 3,8 g/100 ml
  * Osmolarity: 345 mOsm/l
  * Fiber: 1,78 g/100 ml (80% soluble; 20% insoluble).
  Interventions: Dietary Supplement: Diabetes-Specific enteral formula
- Standard Formula (Active Comparator): Standard Enteral Formula:
  * Caloric density: 1,0 kcal/ml
  * Energy: 100 kcal
  * Carbohydrates: 13,8 g/100 ml;
  * Fat: 3,4 g/100 ml
  * Prot: 3,8 g/100 ml
  * Osmolarity: 220 mOsm/l
  * Fiber: 0 g/100 ml
  Interventions: Dietary Supplement: Standard formula

INTERVENTIONS:
Dietary Supplement: Diabetes-Specific enteral formula — Complete enteral formula normocaloric hyperproteic with fiber (80% SOLUBLE)
  Other Names: DIABA
  Arms: Specific Diabetes Formula
Dietary Supplement: Standard formula — Complete enteral formula normocaloric hormoproteic without fiber
  Other Names: Fresubin Original
  Arms: Standard Formula

SUMMARY:
The purpose of this study is to evaluate the effect of a specific nutritional formula for diabetics on the development of hyperglycemia in patients with recent non-diabetic stroke who require admission and enteral nutritional support by nasogastric tube. As well as the effect on metabolic control, development of comorbidities, hospital stay, readmissions, mortality and tolerance of the formula under study.

DETAILED DESCRIPTION:
MAIN GOAL:

To evaluate the effect on the development of hyperglycemia diagnosed as glycemia> 126 mg / dl on an empty stomach or> 150 mg / dl during the infusion of enteral nutrition determined by capillary glycemia during the admission of a specific formula in patients with a first episode of ischemic stroke or hemorrhagic entry into the non-diabetic HCUV stroke unit requiring enteral nutrition by nasogastric tube.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for a first episode of ischemic or hemorrhagic stroke.
* Requiring total enteral nutrition by tube for at least 7 days

Exclusion Criteria:

* Contraindication to enteral nutrition
* Diabetes Mellitus
* Gastrointestinal disease: ulcer, gastritis, diarrhea, gastroparesis, vomiting, abdominal pain
* Need for admission to the ICU
* Previous neurodegenerative disease
* Antibiotherapy for 7 days prior to the inclusion visit
* Allergies or intolerances to any of the components of the formula under study
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
HYPERGLUCEMIA POST-ENTERAL NUTRITION | 2 WEEKS
  Glycemia over 150 mg / dl after the beginning of infusion of complete enteral. nutrition determined by capillary glycemia during admission. Dicotomic variable (Yes/No)

SECONDARY OUTCOMES:
MORTALITY | 3 months
  Mortality during study period. Dicotomic variable (Yes/No)
ORAL FEEDING RECOVERY | 3 months
  Recovery of oral feeding (More than 75% of energy needs) and withdrawal of nasogastric tube during admission. Dicotomic variable (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A De Luis Román, Prof. Dr., Study Director — Service of Endocrinology and Nutrition. Clinic Hospital University of Valladolid; Juan J López-Gómez, Prof. Dr., Principal Investigator — Service of Endocrinology and Nutrition. Clinic Hospital University of Valladolid; Javier F Arenillas-Lara, Prof. Dr., Study Chair — Service of Neurology. Clinic Hospital University of Valladolid
Locations (1):
- Clinic Universitary Hospital, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Gomez JJ, Delgado Garcia E, Primo-Martin D, Simon de la Fuente M, Gomez-Hoyos E, Jimenez-Sahagun R, Torres-Torres B, Ortola-Buigues A, Gomez-Vicente B, Arenillas-Lara JF, De Luis Roman DA. Effect of a diabetes-specific formula in non-diabetic inpatients with stroke: a randomized controlled trial. Nutr Diabetes. 2024 May 30;14(1):34. doi: 10.1038/s41387-024-00292-4. PMID 38816400